CLINICAL TRIAL: NCT05666284
Title: Study of Radiographic Changes and Their Clinical Implications at 2 Years of Implantation of Shortened Uncemented Femoral Stems in Total Hip Arthroplasty
Brief Title: Radiographic Changes and Clinical Implications of Implantation of Shortened Uncemented Femoral Stems in THA
Acronym: THA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8720
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-12

CONDITIONS: Aseptic; Osteonecrosis; Hip Osteoarthritis
Keywords: Hip Osteoarthritis; Aseptic; Osteonecrosis; Coxarthrosis; Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Infertility; Osteonecrosis; Osteoarthritis, Hip; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hip prosthesis market is constantly growing with the number of prostheses reaching 949,000 in 2019. Along with this, there is also an increase in interest in short stems also called shortened stems. Thus on Pubmed, in 5 years, 171 publications have been listed.

Thus, it seems interesting to study and analyze the performance of the shortened stem used in the Department of Orthopedic Surgery and Traumatology of the University Hospitals of Strasbourg and to compare them with the results of the literature.

DETAILED DESCRIPTION:
The objective of this study is to observe the appearance of shortened stem radiological abnormalities at least 2 years postoperatively.

ELIGIBILITY:
Inclusion criteria:

* Male or female (age ≥18 years old)
* Subject operated for first-line THA for an indication of centric hip osteoarthritis (including minor dysplasia and coxa profunda) and aseptic osteonecrosis of the femoral head
* Subject who received a THA between January 2015 and December 2019
* Subject who received an uncemented shortened SCC or SCLA femoral stem
* Radiological data available: pre-operative, immediate post-operative and post-operative at a minimum of 2 years (≥24 months)
* Subject not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Subject having expressed its opposition to the reuse of its data for scientific research purposes.
* Patient operated for inflammatory pathology or major dysplasia, recovery
* Associated fractures or sequelae of fractures
* Patient having presented intraoperative or early complications such as infections, intraoperative fracture, dislocation of the hip following the installation of the THA
* Revision of hip arthroplasty during the study follow-up period for a cause not studied in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient operated for first-line THA for an indication of centric hip osteoarthritis (including minor dysplasia and coxa profunda) and aseptic osteonecrosis of the femoral head
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone changes around the femoral implant at 2 years on hip radiographs. | 2 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique et de Traumatologie du Membre Inférieur - CHU de Strasbourg - France, Strasbourg, France